CLINICAL TRIAL: NCT05217160
Title: Pilot Study: KeraStat® Gel for Topical Delivery of Morphine for Management of Non-Healing, Painful Open Wounds and Ulcers
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Metis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KeraStat
Record Dates: First submitted 2022-01-05; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Wound of Skin; Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either treatment with Kerastat or treatment with Kerastat with Morphine.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, care givers and the investigators will be blinded to which treatment group the participants are randomized to receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- KeraStat® Gel with Morphine (Experimental): Administration and application of KeraStat® Gel with Morphine (Bi-Weekly):
  KeraStat® Gel with Morphine will be formulated by mixing liquid Morphine 25mg/mL into 5mg of KeraStat, this will be individually packaged in 5mL tubes at a concentration of 5mg/mL. Each 5mL tube will cover and area of 300cm2 which is approximately 1.5% TBSA of an average, 60kg subject.
  Home Administration and application of KeraStat® Gel with Morphine (Every 1-3days):
  Dressing is to be changed every 1-3 days, no more than once a day. Subjects will be provided the appropriate amount of pre-compounded KeraStat® Gel with Morphine in 5mL tubes.
  Instructions for application as above will be taught to subjects and instructions will be provided as subjects themselves or designated caretakers or home-care personnel will change their dressings as instructed by their physician with the addition of KeraStat® Gel administration as outlined above.
  Interventions: Drug: KeraStat® Gel with Morphine application
- KeraStat® Gel (Active Comparator): Administration and application of KeraStat® Gel (Bi-Weekly):
  Each 5mL tube will cover and area of 300cm2 which is approximately 1.5% TBSA of an average, 60kg subject.
  Home Administration and application of KeraStat® Gel (Every 1-3days):
  Dressing is to be changed every 1-3 days, no more than once a day. Subjects will be provided the appropriate amount of pre-compounded KeraStat® Gel 5mL tubes.
  Instructions for application as above will be taught to subjects and instructions will be provided as subjects themselves or designated caretakers or home-care personnel will change their dressings as instructed by their physician with the addition of KeraStat® Gel administration as outlined above.
  Interventions: Drug: KeraStat® Gel application

INTERVENTIONS:
Drug: KeraStat® Gel with Morphine application — Administration and application of KeraStat® Gel with Morphine (Bi-Weekly):
  KeraStat® Gel with Morphine will be formulated by mixing liquid Morphine 25mg/mL into 5mg of KeraStat, this will be individually packaged in 5mL tubes at a concentration of 5mg/mL. Each 5mL tube will cover and area of 300cm2 which is approximately 1.5% TBSA of an average, 60kg subject.
  Home Administration and application of KeraStat® Gel with Morphine (Every 1-3days):
  Dressing is to be changed every 1-3 days, no more than once a day. Subjects will be provided the appropriate amount of pre-compounded KeraStat® Gel with Morphine in 5mL tubes.
  Arms: KeraStat® Gel with Morphine
Drug: KeraStat® Gel application — Administration and application of KeraStat® Gel (Bi-Weekly):
  Each 5mL tube will cover and area of 300cm2 which is approximately 1.5% TBSA of an average, 60kg subject.
  Home Administration and application of KeraStat® Gel (Every 1-3days):
  Dressing is to be changed every 1-3 days, no more than once a day. Subjects will be provided the appropriate amount of pre-compounded KeraStat® Gel in 5mL tubes.
  Arms: KeraStat® Gel

SUMMARY:
This study is intended to provide information from subjects who currently have painful, chronically open wounds and assess the pain reduction capacity of KeraStat® Gel with Morphine. In gathering data from subjects who have baseline pain from their chronically open wounds, the investigators can then evaluate the capacity of KeraStat® Gel plus Morphine in reducing the subjects daily pain levels, pain associated with dressing changes, and pain medication consumption.

DETAILED DESCRIPTION:
Chronic wounds pose a serious challenge to wound care professionals, as open and non-healing ulcers are often painful and difficult to treat. Patients are less compliant because of their pain and also run the risk of increased pain medication exposure in treating these wounds. A great deal of healthcare resources are dedicated to the treatment of non-healing open wounds. KeraStat® Gel offers a novel method for the topical delivery of Morphine to manage pain during the treatment of healing these problematic wounds.

Proof of concept work showed that a single treatment application of opioid-loaded keratin hydrogels produced extended analgesia that lasted up to two days in both sensitized and non-sensitized models of pain in rodents. This work then moved the proposed product into a porcine large animal study that showed topical morphine did not delay wound healing or re-epithelization and did not impact dermal thickness or Transforming Growth Factor Beta 1 (TGF1). Additionally, pharmacokinetics assessments showed that topical delivery of morphine to a burn wound resulted in no detectable morphine in animal serum.

KeraStat® Gel is a sterile, non-implantable, water-based gelatinous (hydrogel) wound dressing intended to act as a protective covering in the management of a variety of partial thickness dermal wounds. Keratin is a structural, filamentous protein that, when hydrated, forms a hydrogel that provides coverage and maintains a moist environment for injured skin, similar to collagen and other extracellular matrix molecules used in existing products. Therefore, KeraStat® Gel is expected to behave in an equivalent manner to conventional biopolymer wound dressings. ISO 10993 biocompatibility studies and performance testing, both in vitro and in vivo, indicated that KeraStat® Gel is safe and biocompatible. Additionally, two clinical studies support the assertion that the product is non-sensitizing, non-irritating, and does not produce a humoral response. The current study is designed to provide pilot data to inform a power calculation to determine whether KeraStat® Gel plus Morphine reduces pain associated with dressing changes which may secondarily reduce daily pain and pain medication consumption.

This study is intended to evaluate the efficacy of KeraStat® Gel with Morphine in treating and/or minimizing the pain associated with chronic open wounds and subsequently replace or reduce the need for systemic analgesia.

Long-term impacts include improving tolerance to dressing changes resulting in better adherence to the treatment of painful open wounds, as well as giving providers an alternative to systemic narcotics which are dangerous, have many negative side effects, and are highly addictive. Data from this project will also support further studies in evaluating and assessing patients who have painful wounds and their chronic management.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 18 or older able to provide informed consent.
2. Ulcer size 1-300 cm2

4. Undermining/tunneling <3 cm from wound margin 5. Grossly free of necrotic and/or infected tissue 6. Baseline minimum of 2 on VAS pain scale

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. Known allergy to the standard of care or any of the ingredients in KeraStat® Gel or to morphine
2. Wound has heavy or high-volume exudate or necrotic tissue
3. Clinical signs of infection or contamination of the wound
4. Subjects unable to complete the VAS pain score in pain journal
5. Pregnant or nursing
6. Prisoner
7. Any condition the Investigator determines will compromise subject safety or prevent the subject from completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Scale | Day 0 and Every 2 weeks for up to 12 weeks
  This unidimensional measure is composed of a line, usually 10 centimeters in length, anchored by two verbal descriptors representing the symptom extremes ("no pain" and "worst imaginable pain") and 6 facial expression anchors.
Change in Adverse event assessment | Day 0 and Every 2 weeks for up to 12 weeks
  Assessment of adverse events throughout the course of the subject treatment.

SECONDARY OUTCOMES:
Change in Pressure Sore Quality of Life questionnaire | Day 0 and Every 2 weeks for up to 12 weeks
  Standardized method to assess wound specific symptoms and functional outcomes for quantifying the benefits of associated interventions. The questionnaire is composed of 11 questions with 4 answer boxes for each question, the subject is asked to check one of the four boxes to evaluate the wound. The boxes are labeled No bother at all, A little bother, A lot of bother, and I had this problem but not because of my pressure sores.

CONTACTS AND LOCATIONS:
Locations (1):
- South Texas Aesthetic and Reconstructive Surgery, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No